CLINICAL TRIAL: NCT02200640
Title: A Prospective, Randomized, Double-Blind, Double-Dummy, Titration-to-Response Trial Comparing MICARDIS® (Telmisartan) (40 & 80 mg QD) and COZAAR® (Losartan) (50 & 100 mg QD) in Patients With Mild-to-Moderate Hypertension Using Ambulatory Blood Pressure Monitoring
Brief Title: A Trial Comparing MICARDIS® (Telmisartan) and COZAAR® (Losartan) in Patients With Mild-to-Moderate Hypertension Using Ambulatory Blood Pressure Monitoring (ABPM)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 502.343
Record Dates: First submitted 2014-07-24; First posted 2014-07-25 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2014-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan; Losartan

ARMS (4):
- Low dose of Micardis® (Experimental)
  Interventions: Drug: Low dose of Micardis®, once daily; Drug: Placebo
- High dose of Micardis® (Experimental)
  Interventions: Drug: High dose of Micardis®, once daily; Drug: Placebo
- Low dose of COZAAR® (Active Comparator)
  Interventions: Drug: Low dose of COZAAR®, once daily; Drug: Placebo
- High dose of COZAAR® (Active Comparator)
  Interventions: Drug: High dose of COZAAR®, once daily; Drug: Placebo

INTERVENTIONS:
Drug: High dose of Micardis®, once daily
  Other Names: Telmisartan
  Arms: High dose of Micardis®
Drug: Low dose of Micardis®, once daily
  Other Names: Telmisartan
  Arms: Low dose of Micardis®
Drug: Low dose of COZAAR®, once daily
  Other Names: Losartan
  Arms: Low dose of COZAAR®
Drug: High dose of COZAAR®, once daily
  Other Names: Losartan
  Arms: High dose of COZAAR®
Drug: Placebo

SUMMARY:
The primary aim of the trial is to compare the influence of MICARDIS® (telmisartan 40-80 mg) and COZAAR® (losartan 50-100 mg) in lowering ambulatory diastolic blood pressure (DBP) during the last 6 hours of the 24-hour dosing interval as measured by ABPM after 8-weeks treatment. Secondary objectives include evaluations of: 1) change from baseline in mean systolic blood pressure (SBP) during the last 6 hours of the 24-hour dosing interval as measured by ABPM, 2) changes from baseline in SBP and DBP during other periods during the 24-hour ABPM profile, 3) changes from baseline in mean seated trough SBP and DBP as measured by manual cuff sphygmomanometer, and 4) responder rates based on both ABPM and trough cuff blood pressure

ELIGIBILITY:
Inclusion Criteria:

* Mild-to-moderate hypertension defined as a mean seated diastolic blood pressure of ≥ 95 mmHg and ≤ 109 mmHg, measured by manual cuff sphygmomanometer, on the last visit (Visit 6) of the four-week placebo run-in period (baseline BP). The manual cuff value is calculated as the mean of three seated measurements taken two minutes apart, after the patient has been seated quietly for 5 minutes
* A 24-mean DBP of ≥ 85 mmHg at Visit 7 as measured by ABPM
* Age 18 years or older
* Ability to stop current antihypertensive therapy without risk to the patient (investigator's discretion)
* Ability to provide written informed consent

Exclusion Criteria:

* Pre-menopausal women (last menstruation ≤ 1 year prior to start of run-in period) who:

  * are not surgically sterile; and/or
  * are nursing
  * are of child-bearing potential and are NOT practicing acceptable means of birth control, do NOT plan to continue using this method throughout the study and do NOT agree to submit to periodic pregnancy testing during participation in studies of ≥ 3-months duration. Acceptable methods of birth control include intrauterine device (IUD), oral, implantable or injectable contraceptives
* Mean sitting SBP ≥ 180 mmHg or mean sitting DBP ≥ 110 mmHg during any visit of the placebo run-in period
* Hepatic and/or renal dysfunction as defined by the following laboratory parameters:

  * Serum glutamate-pyruvate-transaminase (alanine aminotransferase) or serum glutamate-oxaloacetate-transaminase (aspartate aminotransferase) greater than two times the upper limit of normal
  * Serum creatinine > 2.3 mg/dL
* Clinically relevant sodium depletion, hyperkalemia, or hypokalemia
* Uncorrected volume depletion
* Primary aldosteronism
* Biliary obstructive disorders
* Known or suspected secondary hypertension
* Hereditary fructose intolerance
* Bilateral renal artery stenosis; renal artery stenosis in a solitary kidney; post-renal transplant patients, presence of only one functioning kidney
* Congestive heart failure (NYHA functional class congestive heart failure (CHF) class III-IV)
* Unstable angina within the past three months
* Stroke within the past six months
* Myocardial infarction or cardiac surgery within the past three months
* Percutaneous transluminal coronary angioplasty (PTCA) within the past three months
* History of angioedema
* Sustained ventricular tachycardia, atrial fibrillation, atrial flutter or other clinically relevant cardiac arrhythmias as determined by the investigator
* Hypertrophic obstructive cardiomyopathy, aortic stenosis, hemodynamically relevant stenosis of the aortic or mitral valve
* Patients with insulin-dependent diabetes mellitus whose diabetes hast not been stable and controlled for at least the past three months as defined by an HbA1c ≥ 10%
* Known drug or alcohol dependency within the past 6 months
* Concomitant administration of medications known to affect blood pressure, except medications allowed by the protocol
* Night shift workers who routinely sleep during the daytime and whose work hours include midnight to 4:00 ante meridien (AM)
* Patients receiving any investigational therapy within one month of signing the informed consent form
* Known hypersensitivity to any component of the formulations
* Any clinical condition which, in the opinion of the investigator would not allow safe completion of the protocol and safe administration of trial medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 333 (Actual)
Dates: Start 2000-03; Primary Completion 2000-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in mean diastolic blood pressure | Up to 8 weeks after start of treatment
  Measured during the last 6 hours of the 24-hour dosing interval using ABPM

SECONDARY OUTCOMES:
Change from baseline in mean systolic blood pressure | Up to 8 weeks after start of treatment
  Measured during the last 6 hours of the 24-hour dosing interval using ABPM
Changes from baseline in diastolic and systolic blood pressure | Up to 8 weeks after start of treatment
  Measured during other times of the 24-hour ABPM profile (e.g. 24-hour mean, morning mean, daytime mean and nighttime mean)
Changes from baseline in mean seated trough diastolic blood pressure and systolic blood pressure | Up to 8 weeks after start of treatment
  Triplicate measurement in two minute intervals after 5 minutes of rest, in seated position using sphygmomanometer
Assessment of responder rates on ABPM | Baseline, 8 weeks after start of treatment
Assessment of responder rates on trough cuff blood pressure | Baseline up to 8 weeks after start of treatment